CLINICAL TRIAL: NCT02772588
Title: ARN-509+Abiraterone Acetate+Leuprolide With Stereotactic, Ultra-Hypofractionated Radiation (AASUR) in Very High Risk Prostate Cancer: A Single Arm, Phase II Study
Brief Title: AASUR in High Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Weill Medical College of Cornell University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-334; c15-164 (Other: Prostate Cancer Clinical Trials Consortium, LLC (PCCTC))
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: ARN-509; Abiraterone; Leuprolide; Intensity-Modulated and Image-Guided Radiation Therapy; 15-334; apalutamide,; JNJ-56021927
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; abiraterone; Leuprolide

ARMS (1):
- patients with prostate cancer (Experimental): Eligible patients will receive a total of 6 months of leuprolide, abiraterone, and ARN-509 to begin three months prior to RT and continuing until approximately 3 months post-RT. Patients will be assessed every 4 weeks (±1 week) (a cycle = 28 days) throughout their treatment with the study drugs, and at least once during RT.
  Interventions: Drug: ARN-509; Drug: Abiraterone; Drug: Leuprolide; Radiation: stereotactic, ultra-fractionated radiotherapy

INTERVENTIONS:
Drug: ARN-509
  Other Names: apalutamide; JNJ-56021927
Drug: Abiraterone
Drug: Leuprolide
Radiation: stereotactic, ultra-fractionated radiotherapy

SUMMARY:
The purpose of this study is to determine whether anti-testosterone medications, when administered before, during, and after high-dose, precision radiation, will be effective in preventing the prostate cancer from returning.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologic evidence of adenocarcinoma of the prostate confirmed at local institution.
* At least one of the following:
* Two or more high risk features OR
* Gleason score 8-10
* PSA ≥20 ng/mL within two months prior to registration
* Clinical Stage ≥T3 disease, as determined by standard digital rectal examination (DRE)
* Radiographic stage ≥T3 disease as determined by a ≥75% probability of extracapsular extension or seminal vesicle invasion per reading radiologist
* Any Gleason 9 or 10 disease OR >4 cores of Gleason 8 disease
* KPS ≥ 70%
* IPSS (International Prostate Symptom Score) ≤ 20F
* Patient must be available for follow-up
* Laboratory test findings within 28 days of study registration :
* Adequate hepatic function:
* Bilirubin ≤ 1.5 times the upper institutional limits of normal (ULN). Patients with a history of Gilbert's syndrome may be enrolled if the total bilirubin is < 3 mg/dL with a predominance of indirect bilirubin. If the total bilirubin is >1.5 x the institutional ULN, direct and indirect bilirubin will be measured and if direct bilirubin is ≤ 1.5 x the institutional ULN, the patient will be eligible to participate
* SGPT (ALT) and SGOT (AST) ≤ 2.5 x ULN
* Adequate renal function with creatinine <2.0 x the institutional ULN
* Adequate hematologic function:
* Absolute neutrophil counts ≥ 1500 cell/mm3
* Platelets ≥ 100,000 cells/mm3 (independent of blood transfusion and/or growth factors within 3 months prior to registration)
* Hemoglobin value ≥9 g/dL at the Screening Visit (independent of blood transfusion and/or growth factors within 3 months prior to registration)
* Albumin ≥ 3.0 g/dL
* Potassium ≥ 3.5 mmol/L
* Patients with pelvic and/or retroperitoneal lymph nodes < 1.5 cm in short axis are eligible as they are not considered to have definitive metastases
* Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information NOTE: HIPAA authorization may be either included in the informed consent or obtained separately
* Males 18 years of age and above
* The effects of apalutamide, abiraterone, leuprolide and stereotactic, ultra-hypofractionated radiation on the developing human fetus at the recommended therapeutic dose are unknown. Men (including men with vasectomies) must agree to use adequate contraception (a condom and another effective method of birth control) prior to registration, for the duration of study participation, and for at least 3 months thereafter. Men must also agree not to donate sperm for the duration of study participation, and for at least 3 months thereafter.

Exclusion Criteria:

* Radiographic evidence of metastatic disease
* Patients with one or more positive lymph nodes as determined by radiographic assessment of MRI or CT NOTE: lymph nodes noted on MRI or CT to be > 1.5 cm on the short axis will require review by the local reference radiologist per institutional RECIST review practices. If the lymph nodes are considered suspicious on repeat review, they must be confirmed negative for study participation
* Prior treatment for prostate cancer; this includes any prior surgery (including Transurethral resection of the prostate (TURP), prostate cancer treatment), chemotherapy, radiation, or anti-androgen therapy/androgen deprivation therapy with the following exception: patients who will have been on LHRH Agonist/Antagonist Therapy for </= 1 month prior to registration are permitted to enroll with study PI approval.
* Prior use of steroidal antiandrogens (megestrol acetate, cyproterone acetate), AR partial agonists, ketoconazole, chemotherapy, immunotherapy, estrogens, radiopharmaceuticals within 3 months before registration
* Prior use of non-steroidal anti-androgens (e.g., bicalutamide, flutamide, nilutamide) within 1 month before registration
* Prior treatment with medications known to lower the seizure threshold within 4 weeks of registration (see section 5.5.2 apalutamide for a list of prohibited medications)
* History of another malignancy within the previous 3 years except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, adequately treated Stage I or Stage II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 3 years
* Severe hepatic impairment (Child-Pugh Class C)
* Concurrent treatment with strong CYP3A4 inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital)
* Major surgery within 4 weeks of registration
* Presence of a pacemaker
* Active infection or other medical condition that would make prednisone use contraindicated
* A known hypersensitivity to abiraterone acetate, apalutamide, and prednisone and/or any of their excipients
* Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to registration.
* Seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
* Any ECG changes that interfere with QT interval interpretation (e.g., left bundle branch block, frequent premature ventricular contractions)
* Prolonged QTc >450ms at the Screening Visit
* Uncontrolled diabetes, heart disease, hypertension
* Gastrointestinal disorder that may affect absorption of study treatment
* Active symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Active Infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis) or other medical condition that would make prednisone/prednisolone corticosteroid) use contraindicated
* Patients with Crohn's disease or ulcerative colitis
* Patients that cannot tolerate MRI
* Inability to have fiducial markers placed
* Any condition that in the opinion of the investigator, would preclude participation in this study
* Enrollment concurrently in another investigational drug study or within 4 weeks of registration
* Concurrent treatment with strong CYP3A4 inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
proportion of patients with biochemical failure | 36 months
  Biochemical failure is defined as an increase in PSA by more than 2ng/mL above the nadir value. PSA rise equals or exceeds 2ng/mL will be the date of failure.

CONTACTS AND LOCATIONS:
Overall Officials: Sean M McBride, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - John Hopkins Medical Center, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Rockville, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/